CLINICAL TRIAL: NCT02999490
Title: 18F-FDG PET/CT in Diagnostic Patients of Disorder of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Jing Zhao, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYXK0001
Record Dates: First submitted 2016-03-25; First posted 2016-12-21 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Persistent Vegetative State
MeSH Terms: conditions — Persistent Vegetative State | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controls (No Intervention): The controls are intravenous injected of 185 to 370 MBq 18F-FDG.Then,the controls sleep for an hour in a quiet room before scanning.
- Patients (Experimental): The patients are intravenous injected of 185 to 370 MBq 18F-FDG.Then,the patients sleep for an hour in a quiet room before scanning.
  Interventions: Radiation: 18F-FDG

INTERVENTIONS:
Radiation: 18F-FDG — 18F-FDG is positron emission tomography imaging agent which is already widely used in PET/CT examination.
  Arms: Patients

SUMMARY:
Clinical examinations are difficult to discriminate between vegetative state and minimally conscious state. the diagnostic and prognostic usefulness of neuroimaging methods has not been established in a clinical setting. we will do a forward study of PET imaging in disorders of consciousness patients, and validate with clinical assessments with the coma recovery Scale-Revised(CRS-R).

DETAILED DESCRIPTION:
Every patient need to be conducted the PET/CT scanning two times.The first time is resting state.The second time is stimulated state by watching a vedio.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of disorder of consciousness

Exclusion Criteria:

-

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
standardized uptake value | 60 mins after injecting 18F-FDG

CONTACTS AND LOCATIONS:
Overall Officials: Yin Jilin, Study Director
Locations (1):
- The PET/CT Centre Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes